CLINICAL TRIAL: NCT06457581
Title: Effectiveness of Dry Needling Adjuvant to Selective Serotonin Reputake Inhibitors Versus Trigger Point Injection for Pain Management in Fibromyalgia
Brief Title: Effectiveness of Dry Needling Adjuvant to Selective Serotonin Reputake Inhibitors vs TP Injection for Pain Management
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/724
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Pain; Fibromyalgia
MeSH Terms: conditions — Pain; Fibromyalgia | interventions — Dry Needling; Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling (Other)
  Interventions: Other: Dry Needling; Drug: serotonin reuptake inhibitor (SSRI)
- Trigger points injections (Experimental)
  Interventions: Procedure: Trigger points injections

INTERVENTIONS:
Other: Dry Needling — Group A will undergo dry needling sessions twice a week over eight weeks, specifically targeting trigger points and tender points. Simultaneously, a consistent dosage of selective serotonin reuptake inhibitor (SSRI) will be administered and maintained throughout the entire duration of the study.
  Arms: Dry Needling
Procedure: Trigger points injections — Group B will undergo a comprehensive intervention involving trigger point injections administered biweekly over eight weeks. These injections will specifically target trigger points. Additionally, a control measure will be implemented through simulated needling at non-specific points.
  Arms: Trigger points injections
Drug: serotonin reuptake inhibitor (SSRI) — serotonin reuptake inhibitor (SSRI)
  Arms: Dry Needling

SUMMARY:
The principal objective is to contribute valuable insights that hold direct implications for medical practice and patient care, with the potential to influence health policy pertaining to fibromyalgia management.

DETAILED DESCRIPTION:
The study aims to outline distinct patient subgroups manifesting heightened responsiveness to one therapeutic intervention vis-à-vis the other, thereby facilitating the formulation of more personalized and efficacious treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

* Stable on SSRIs for at least three months (for Group A)
* Age between 18 and 65 years
* Participants suffering from recent cervical pain without any pathology

Exclusion Criteria:

* Presence of any other chronic pain conditions.
* Contraindications to SSRIs or trigger point injections.
* Pregnancy or lactation.
* History of psychiatric disorders other than depression and anxiety

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | 12 Months
  It includes 19 items that generate seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The total score ranges from 0 to 21, with higher scores indicating poorer sleep quality.
Fibromyalgia Impact Questionnaire: | 12 months
  It includes questions related to physical functioning, work status, depression, anxiety, sleep, pain, stiffness, fatigue, and well-being. Scores on the FIQ range from 0 to 100, with higher scores indicating greater impact and symptom severity

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudary Muhammad Akram Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No